CLINICAL TRIAL: NCT03735173
Title: Randomized Clinical Trial Comparing the Outcome of Cemented All-Polyethylene Pegged vs. Keeled Components Through a Subscapularis Tenotomy or a Subscapularis Peel
Brief Title: Comparing the Outcome of Cemented All-Polyethylene Pegged vs. Keeled Components Through a Subscapularis Tenotomy or a Subscapularis Peel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark E. Morrey, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-011251
Record Dates: First submitted 2018-10-04; First posted 2018-11-08 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Arthropathy Shoulder; Shoulder Pain; Shoulder Osteoarthritis; Shoulder Arthritis; Shoulder Arthropathy Associated With Other Conditions; Necrosis of Bone; Arthritis; Inflammatory Arthritis
MeSH Terms: conditions — Shoulder Pain; Osteonecrosis; Arthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Pegged through SP (Active Comparator): Primary anatomic shoulder arthroplasty with implantation of a cemented all-polyethylene pegged glenoid component through a Subscapularis Peel (SP) manipulation.
  Interventions: Procedure: ReUnion TSA, pegged design
- Pegged through ST (Active Comparator): Primary anatomic shoulder arthroplasty with implantation of a cemented all-polyethylene pegged glenoid component through subscapularis tenotomy (ST) manipulation.
  Interventions: Procedure: ReUnion TSA, pegged design
- Keeled through SP (Active Comparator): Primary anatomic shoulder arthroplasty with implantation of a cemented all-polyethylene keeled glenoid component through a Subscapularis Peel (SP) manipulation.
  Interventions: Procedure: ReUnion TSA, keeled design
- Keeled through ST (Active Comparator): Primary anatomic shoulder arthroplasty with implantation of a cemented all-polyethylene keeled glenoid component through subscapularis tenotomy (ST) manipulation.
  Interventions: Procedure: ReUnion TSA, keeled design

INTERVENTIONS:
Procedure: ReUnion TSA, pegged design — ReUnion total shoulder arthroplasty system, pegged design
  Arms: Pegged through SP; Pegged through ST
Procedure: ReUnion TSA, keeled design — ReUnion total shoulder arthroplasty system, keeled design
  Arms: Keeled through SP; Keeled through ST

SUMMARY:
Participants who choose to participate in this study, will either have their tendon repaired to tendon, so-called tenotomy repair, or tendon repaired to bone, so-called peel repair.

ELIGIBILITY:
Inclusion Criteria:

* Subjects willing to sign the informed consent
* Male and female subjects ages 18 - 90 at the time of surgery
* Subjects indicated for an anatomic total shoulder arthroplasty (including primary glenohumeral osteoarthritis, avascular necrosis, and inflammatory arthritis)

Exclusion Criteria:

* Inability to comply with follow-up requirements
* Known or presumed substantial rotator cuff disorders
* Subjects with an active or suspected latent infection in or about the shoulder
* Subjects with instability (surgically or non-surgically addressed)
* Subjects presenting with posttraumatic avascular necrosis
* Need for glenoid bone grafting
* Pregnant subjects

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Function of Subscapularis muscle as measured by belly-press test | 5 years
Radiographic loosening | 5 years
  "glenoid at risk" proportion

CONTACTS AND LOCATIONS:
Overall Officials: Mark Morrey, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials